CLINICAL TRIAL: NCT07280143
Title: The Development of MASLD Among Survivors of Breast or Colorectal Cancer
Acronym: EVALUATE
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: EVALUATE; DRKS00038398 (Registry Identifier: DRKS)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Survivors; Colorectal (Colon or Rectal) Cancer Survivors; MASLD/MASH (Metabolic Dysfunction-Associated Steatotic Liver Disease / Metabolic Dysfunction-Associated Steatohepatitis)
Keywords: MASLD; Cancer survivorship; Survivorship care; Non-invasive imaging; Liver fibrosis screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer survivors
- Colorectal cancer survivors

SUMMARY:
A metabolic issue is a condition where the body has problems with converting food into energy, using energy or storing energy properly. Examples of metabolic issues include obesity, diabetes, or high blood pressure

MASLD -Metabolic-associated steatotic liver disease - also known as non-alcoholic fatty liver disease, is a condition where fat builds up in the liver due to metabolic issues. Excess liver fat can cause inflammation, scaring, also known as fibrosis, and over time, lead to liver failure.

MASLD can have different severities. Non-fibrotic MASLD is when there is a small amount of fat in the liver and usually does not cause major problems. However, it can get worse over time and can develop into fibrotic MASLD.

MASLD is very common, about one-third of the world's population is affected. In Switzerland, it is predicted that one-quarter of the Swiss population is affected by it. MASLD can affect anyone who has any metabolic issues, however it seems like some medications, such as cancer treatments, could play a role in MASLD development.

Studying MASLD is important because it is very common. Learning more about it can help doctors find better ways to diagnose and treat the condition.

Furthermore, it is important to find out who would be more likely to develop MASLD. People who are more likely could maybe do some regular testing to diagnose it early and start treatment before it is worsening. Early diagnosis is important since liver damage can be reversed with lifestyle changes, diet or medication.

Cancer survivors are at a higher risk of developing MASLD due to changes in their metabolism, lifestyle as well as side effects of cancer treatments. However, MASLD is often underdiagnosed in cancer survivors, even though it can increase the risk of future health complications.

Currently, liver biopsy is the standard method of diagnosing MASLD, as it provides the most accurate results. However, liver biopsy is uncomfortable and carries risks like pain and infections.

Newer non-invasive technologies, such as ultrasound-based vibration-controlled transient elastography (VCTE, also known as FibroScan®) and Magnetic Resonance Imaging (MRI), show promise in detecting liver fibrosis earlier and more safely. However, they are not yet widely used because they are not as precise as biopsy at detecting liver inflammation.

EVALUATE is an observational study performed by the Department of Clinical Research at the University of Bern. In collaboration with the Department of Hepatology, Inselspital, University Hospital of Bern and the Department of Radiology, University Cancer Centre Inselspital.

EVALUATE will use two of the newer, less painful methods - VCTE and MRI to check for signs of fibrotic MASLD. Combined with a blood test, a score can be calculated to see if someone is at high-risk for advanced MASLD.

In the case that the results from the main study are uncertain, the participant will be asked to participate in an MRI sub study.

This study will help improve ways to check for liver disease in cancer survivors, leading to early detection and quicker treatment. Eventually the information of this study could help create better guidelines and improve care for cancer survivors at risk of liver problems.

ELIGIBILITY:
Inclusion criteria:

* Signed Informed consent form
* Age ≥ 18 years
* Diagnosis of BC or CRC at least 5 years but no more than 10 years before enrollment, and no recurrence or new cancer diagnoses during this time period (except for superficial non-melanoma skin cancer or superficial bladder cancer or cancer in-situ). Patients who received/are still receiving adjuvant therapy may be included. Time period is calculated from date of first histological diagnosis of cancer.

Exclusion criteria:

* Known or suspected chronic hepatic disease
* Pregnancy, or suspected pregnancy (as liver stiffness and fat content are often elevated but reverse after childbirth)
* For the MRI sub-study: Contraindication to MRI, including: claustrophobia and presence of metal implants or devices or foreign metal objects in/on the body, such as pacemakers, defibrillators, prosthetic cardiac valves, cochlear implants, metal clips e.g., vascular clips, spinal cord stimulators or deep brain stimulators, shrapnel or bullet fragments, metal in the eyes, orthopedic hardware and piercings that cannot be easily removed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast and colorectal cancer survivors
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-07-14 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
High probability of fMASLD | Month 3
  Description:
  Dichotomous measure (Yes/No) of high probability of fibrotic MASLD (fMASLD) based on FAST and MAST score thresholds:
  * Yes if the FAST score indicates high probability (FAST ≥ 0.67), or
  * Yes if the FAST score indicates uncertain probability (FAST > 0.35 and < 0.67) and the MAST score indicates high probability (MAST ≥ 0.242).
  * No otherwise.
  Unit of Measure:
  Yes/No

SECONDARY OUTCOMES:
Participant age | Day 1 (at enrollment)
  Age of the participant at the time of enrollment, recorded in years.
  Unit of Measure:
  Years
Participant sex | Day 1 (at enrollment)
  Sex of the participant recorded at the time of enrollment (male or female).
  Unit of Measure:
  Categorical (male/female)
Body Mass Index (BMI) | Day 1 (at enrollment)
  Body mass index (BMI) of the participant at the time of enrollment, calculated as weight in kilograms divided by height in meters squared (kg/m²).
  Unit of Measure:
  kg/m²
A Body Shape Index (ABSI) | Day 1 (at enrollment)
  A Body Shape Index (ABSI) of the participant at the time of enrollment, calculated using waist circumference, weight, and height to provide a normalized measure of body shape independent of BMI.
  Unit of Measure:
  Unitless
Waist Circumference | Day 1 (at enrollment)
  Waist circumference of the participant at the time of enrollment, measured in centimeters at the midpoint between the lowest rib and the iliac crest.
  Unit of Measure:
  Centimeters (cm)
Cancer histology | Day 1 (at enrollment)
  Histological classification of the participant's cancer type, determined from biopsy or surgical specimen according to standard pathological criteria.
  Unit of Measure:
  Categorical for breast cancer: for breast cancer:
  * Ductal carcinoma in situ (DCIS)
  * Invasive breast cancer (IDC/ILC)
  * Tripple negative breast cancer (TNBC)
  * Inflammatory breast cancer
  * Other
  Categorical for colorectal cancer:
  Adenocarinoma other
Cancer stage | Day 1 (at enrollment)
  Stage of the participant's cancer at enrollment, determined using standard clinical or pathological staging criteria (e.g., TNM classification or other recognized staging system).
  Unit of Measure:
  Categorical (e.g., Stage I, II, III, IV)
Cancer treatment Received | Day 1 (at enrollment)
  Type of treatment the participant is receiving at enrollment or during the study, categorized by modality (e.g., surgery, chemotherapy, radiation, immunotherapy, or combination therapy).
  Unit of Measure:
  Categorical (e.g., Chemotherapy, Targeted therapy, Hormone therapy, Immunotherapy, Radiation, Supportive or adjunct therapy)
Number of Treatment Cycles | Day 1 (at enrollment)
  Number of treatment cycles received by the participant, recorded as the total count of completed cycles of the assigned therapy at the time of assessment.
  Unit of Measure:
  Count (number of cycles)
Intervals Between Treatment Cycles | Day 1 (at enrollment)
  Time intervals between consecutive treatment cycles for the participant, measured in days from the end of one cycle to the start of the next.
  Unit of Measure:
  Days
Liver Stiffness Measurement (LSM) | Month 3
  Liver stiffness measurement (LSM) of the participant, obtained using elastography or other validated imaging techniques, reported in kilopascals (kPa). LSM provides a quantitative assessment of liver fibrosis and can be used to monitor disease progression or response to treatment.
  Unit of Measure:
  Kilopascals (kPa)
Controlled Attenuation Parameter (CAP) | Month 3
  Controlled Attenuation Parameter (CAP) measured via elastography, reported in decibels per meter (dB/m). CAP provides a quantitative assessment of liver steatosis and can be used to monitor disease severity or response to treatment.
  Unit of Measure:
  Decibels per meter (dB/m)
MRI-Based Liver Stiffness Measurement (MRI-LSM) | Month 3
  Liver stiffness measured using magnetic resonance imaging (MRI-LSM), reported in kilopascals (kPa). MRI-LSM provides a non-invasive quantitative assessment of liver fibrosis and can be used to monitor disease progression or response to therapy.
  Unit of Measure:
  Kilopascals (kPa)
Proton Density Fat Fraction (PDFF) | Month 3
  Proton Density Fat Fraction (PDFF) of the liver measured using MRI, reported as a percentage (%). PDFF provides a quantitative assessment of liver fat content and can be used to monitor liver steatosis and response to intervention.
  Unit of Measure:
  Percent (%)
Agile 3+ Score | Month 3
  Agile 3+ is a composite, non-invasive score used to estimate the probability of advanced liver fibrosis (F3 or higher). It integrates clinical, laboratory, and imaging parameters to provide a continuous or categorical assessment of fibrosis severity, allowing monitoring of disease progression or response to therapy.
  Unit of Measure:
  Continuous score (unitless)
Agile 4 Score | Month 3
  Agile 4 is a composite, non-invasive score used to estimate the probability of cirrhosis or very advanced liver fibrosis (F4). It combines clinical, laboratory, and imaging parameters to provide a continuous or categorical assessment, allowing monitoring of disease progression or response to therapy.
  Unit of Measure:
  Continuous score (unitless)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Segelov, Prof., Principal Investigator — Department of Clinical Research, University of Bern
Locations (1):
- Department of Clinical Research, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study website — https://dcr.unibe.ch/research/evaluate_study/index_eng.html